CLINICAL TRIAL: NCT03909373
Title: Validation of the Patient-Specific Functional Survey in Patients With Carpal Tunnel
Brief Title: Validation of PSFS in Carpal Tunnel Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Logistics (Research Staffing)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Other Study IDs: 49525
Record Dates: First submitted 2019-03-07; First posted 2019-04-10 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: patients with carpal tunnel syndrome
  Interventions: Other: PSFS

INTERVENTIONS:
Other: PSFS — Patients will complete the patient specific functional scale. no intervention being administered

SUMMARY:
Validation of the Patient Specific Functional Scale in patients with carpal tunnel syndrome

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of carpal tunnel syndrome

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Principal Investigator who meet inclusion criteria
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Specific Functional Scale Scores | 2 weeks after initial completion
  PSFS measures perceived function. Patients rate their ability to perform self-selected tasks on a 0-10 scale, with higher scores indicating higher ability.
Patient Specific Functional Scale Scores | 6 weeks after surgery
  Patients rate their ability to perform self-selected tasks on a 0-10 scale, with higher scores indicating higher ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD